CLINICAL TRIAL: NCT04050254
Title: Effects of Transcranial Direct Current Stimulation Combined With Therapeutic Exercise in Fibromyalgia Patients. A Triple-blinded, Randomized, Placebo-controlled Trial
Brief Title: tDCS Combined With Therapeutic Exercise in Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: tDCS+ET-Fibromyalgia
Record Dates: First submitted 2019-06-14; First posted 2019-08-08 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Fibromyalgia
Keywords: tDCS; Therapeutic exercise; Referred pain; Central sensitization
MeSH Terms: conditions — Fibromyalgia; Pain, Referred | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Real tDCS + exercise (Experimental): Transcranial direct current stimulation combined with therapeutic exercise
  Interventions: Device: Real tDCS; Device: Therapeutic exercise
- Sham tDCS + exercise (Sham Comparator): Sham transcranial direct current stimulation combined with therapeutic exercise
  Interventions: Device: Sham tDCS; Device: Therapeutic exercise
- Control (No Intervention): No treatment.

INTERVENTIONS:
Device: Real tDCS — Real tDCS (STARTSTIM® 8 stimulator, Neuroelectric Barcelona, Spain) for five sessions on alternate days.tDCS is a galvanic current applied by a cap for 20 minutes at an intensity of 2 milliamps.
  Arms: Real tDCS + exercise
Device: Sham tDCS — Sham current (STARSTIM® 8 stimulator, Neuroelectric Barcelona, Spain) for five sessions on alternate days. Sham tDCS will be applied for the same time than real tDCS.
  Arms: Sham tDCS + exercise
Device: Therapeutic exercise — The therapeutic exercise program will include aerobic exercise and muscle strengthening for five sessions on alternate days. The program will include exercises and will last 30-45 minutes.
  Arms: Real tDCS + exercise; Sham tDCS + exercise

SUMMARY:
The purpose of this study is to assess the effects on pain of transcranial direct current stimulation combined with therapeutic exercise in fibromyalgia patients.

DETAILED DESCRIPTION:
Fibromyalgia is one of the rheumatic diseases with the greatest impact on the quality of life, whose etiology and pathophysiology is not yet fully demonstrated. Perhaps this is why its therapeutic approach is refractory to current treatments.

Based on the theory that fibromyalgia is characterized by a sensitization at the level of the central nervous system that leads to an increase in the perception of pain, any therapeutic approach aimed at modulating the central nervous system may be beneficial. Electrical stimulation with transcranial direct current (tDCS) is among these techniques.

In the same way, therapeutic exercise has shown to have, like the tDCS, a beneficial effect on pain in different chronic pathologies.

The present study aims to investigate the effect on pain of a combination therapy of tDCS and therapeutic exercise in patients with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Fulfilled the 2010 American Colleague of Rheumatology criteria for fibromyalgia.
* Normal pain intensity of 4 or more points on a visual analog scale.
* Able to participated in a therapeutic exercise program.
* Understanding of spoken and written Spanish.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Metallic implants in the head.
* Tumor, trauma or surgery in the brain.
* Epilepsy or stroke.
* History of substance abuse in the last 6 months.
* Use of carbamazepine in the last 6 months.
* Severe depression (Beck Depression Index II of 29 or more).
* Diagnosed psychiatric pathology.
* Rheumatic pathology not medically controlled.
* Coexisting autoimmune pathology.
* Chronic inflammatory disease (rheumatoid arthritis, erythematosus systemic lupus, inflammatory bowel disease).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2020-03-27 (Actual)

PRIMARY OUTCOMES:
Change in referred pain area after suprathreshold pressure stimulation from baseline to post-treatment | Baseline; immediately after intervention; 1-month after intervention
  A pressure algometer (Force Ten™, Wagner Instruments, USA) will be used. It will be performed on the infraspinatus muscle (point equidistant between the midpoint of the spine of the scapula, the inferior angle of the scapula and the midpoint of the medial border of the scapula) at a constant suprathreshold pressure (20% above the pressure pain threshold) for 60 seconds.
  After the stimulation, the subject should draw the induced pain area on a digital bodychart using the Navigate Pain application (Navigate Pain, Aalborg University, Denmark).
Change in pain intensity from baseline to post-treatment | Baseline; immediately after intervention; 1-month after intervention
  It will be measured with a visual analog scale (VAS) of 100 millimeters in length. The subject has to indicate the level of pain he feels, being 0 the absence of pain and 100 the maximum imaginable

SECONDARY OUTCOMES:
Fibromyalgia Impact Quality-of-Life | Baseline; immediately after intervention; 1-month after intervention
  It will be measured with the version adapted to the Spanish of the Fibromyalgia Impact Questionnaire (FIQ). The scale ranges from 0 to 100. Higher values represent a worse result.
Anxiety | Baseline; immediately after intervention; 1-month after intervention
  The version adapted to Spanish from the State Scale (STAI-ES) of the State-Trait Anxiety Inventory (STAI) will be used. The scale ranges from 0 to 60. Higher values represent a worse result.
Pain catastrophizing | Baseline; immediately after intervention; 1-month after intervention
  The Spanish version of the Pain Catastrophizing Scale (PCS) will be used. The scale ranges from 0 to 52. Higher values represent a worse result.
Depression | Baseline; immediately after intervention; 1-month after intervention
  The adaptation to the Spanish of Beck Depression Inventory II will be used. The scale ranges from 0 to 63. Higher values represent a worse result.

OTHER OUTCOMES:
Blinding | Immediately after intervention
  Blinding of subjects and researchers will be assessed using the James Index.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Nuestra Señora del Prado, Talavera de la Reina, Toledo, Spain

REFERENCES:
- [Derived] Arroyo-Fernandez R, Avendano-Coy J, Velasco-Velasco R, Palomo-Carrion R, Bravo-Esteban E, Ferri-Morales A. Effectiveness of Transcranial Direct Current Stimulation Combined With Exercising in People With Fibromyalgia: A Randomized Sham-Controlled Clinical Trial. Arch Phys Med Rehabil. 2022 Aug;103(8):1524-1532. doi: 10.1016/j.apmr.2022.02.020. Epub 2022 Mar 22. PMID 35331718